CLINICAL TRIAL: NCT04786119
Title: A Prospective, Multi-center, Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in Unicondylar Knee Arthroplasty (UKA) and Total Knee Arthroplasty (TKA) Procedures
Brief Title: Study to Evaluate the Safety and Effectiveness of REAL INTELLIGENCE™ CORI™ in Knee Arthroplasty Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORI.2019.07
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-09

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Unicompartmental Knee Arthroplasty; Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CORI Robotics (Experimental): Subjects having robotic assisted knee arthroplasty as decided by their doctor and treated with CORI Robotics.
  Interventions: Device: CORI Robotics

INTERVENTIONS:
Device: CORI Robotics — Knee arthroplasty with robotics assisted surgery using the CORI Robotics System.

SUMMARY:
Background: REAL INTELLIGENCE™ CORI™ (CORI Robotics) is a computer-assisted orthopaedic surgical navigation and burring system. CORI Robotics is designed to help surgeons in planning and executing certain types of knee surgery involving bone preparation. These types of surgery are called 'unicondylar knee arthroplasty' (UKA) and 'total knee arthroplasty' (TKA).

Purpose:

This study is being carried out to demonstrate the safety and effectiveness of the CORI Robotics. The data collected will be used to meet the post-market clinical follow-up requirement in Europe and to support claims and publications.

Objectives:

The primary objective of this study is to evaluate the use of CORI Robotics in UKA and TKA procedures in achieving post-operative leg alignment to check that the results of the operation are similar to what the surgeon originally planned.

Research participants / locations:

Research participants will be recruited from up to 8 sites in 4 countries globally (UK, US, Germany and India).

ELIGIBILITY:
Inclusion Criteria:

* The subject's treating clinician has decided that REAL INTELLIGENCE™ CORI™ and a compatible Smith+Nephew Knee Implant System is the best treatment for the subject's unicondylar knee arthroplasty (UKA) or total knee arthroplasty (TKA) and the subject has agreed to the treatment.
* Subject requires a cemented UKA or TKA as a primary indication that meets either criterion A or B.

  * A. Subject requires a cemented UKA as a primary indication due to any of the following conditions:

    1. Non-inflammatory degenerative joint disease, including osteoarthritis
    2. Avascular necrosis
    3. Requires correction of functional deformity
    4. Requires treatment of fractures that were unmanageable using other techniques
  * B. Subject requires a cemented TKA as a primary indication due to any of the following condition:

    1. Degenerative joint disease, including osteoarthritis
    2. Rheumatoid arthritis
    3. Avascular necrosis
    4. Requires correction of functional deformity
    5. Requires treatment of fractures that were unmanageable using other techniques
* Subject is of legal age to consent and considered skeletally mature (≥ 18 years of age at the time of surgery)
* Subject agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the Ethical Committee (EC) or Institutional Review Board (IRB) approved informed consent form.
* Subject plans to be available through one (1) year postoperative follow-up.
* Routine radiographic assessment is possible.
* Subject able to follow instructions and deemed capable of completing all study questionnaires.

Exclusion Criteria:

* Subject receives a CORI Robotics UKA or TKA on the index joint as a revision for a previously failed surgery, or need for complex implants, or any other implant than a standard UKA or TKA (e.g. stems, augments, or custom made devices).
* Subject has been diagnosed with post-traumatic arthritis
* Subject receives bilateral UKA or TKA
* Subject does not understand the language used in the Informed Consent Form.
* Subject does not meet the indication or is contraindicated for UKA or TKA according to specific Smith+Nephew knee system's Instructions For Use (IFU).
* Subject has active infection or sepsis (treated or untreated).
* Subject is morbidly obese with a body mass index (BMI) greater than 40.
* Subject is pregnant or breast feeding at the time of surgery.
* Subject, in the opinion of the Investigator, has advanced osteoarthritis or joint disease at the time of surgery and was better suited for an alternate procedure.
* Subject has a condition(s) that may interfere with the TKA or UKA survival or outcome (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease, or an active, local infection).
* Subject in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
* Subject, in the opinion of the Investigator, has a neuromuscular disorder that prohibited control of the index joint.
* Subject is a prisoner or meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha O'Neill, Study Chair — Smith & Nephew, Inc.
Locations (8):
- United States (4):
  - Orthopedic Institute of the West, Phoenix, Arizona
  - Duke Health, Morrisville, North Carolina
  - OrthoNeuro, New Albany, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Germany (2):
  - Orthopaedic clinic of the Medical School Hannover, Hanover
  - Pius-Hospital Oldenburg, Oldenburg
- Lokmanya Hospital, Pune, Maharashtra, India
- The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited across 8 sites in Europe, United Kingdom, India, and the United States.
Units Other Than Participants: knees
Groups:
- CORI™ in Unicondylar Knee Arthroplasty (UKA): Participants having robotic assisted unicondylar knee arthroplasty (UKA) as decided by their doctor and treated with CORI™ Robotics.
  CORI™ Robotics: UKA with robotics assisted surgery using the CORI™ Robotics System.
- CORI™ in Total Knee Arthroplasty (TKA): Participants having robotic assisted total knee arthroplasty (TKA) as decided by their doctor and treated with CORI™ Robotics.
  CORI™ Robotics: TKA with robotics assisted surgery using the CORI™ Robotics System.
Period: Overall Study
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Started (Number of participants that started the study for the final analysis reporting period) | 55; 55 knees | 71; 71 knees
Completed (Number of participants that completed the study for the final analysis reporting period) | 45; 45 knees | 61; 61 knees
Not Completed | 10; 10 knees | 10; 10 knees
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 5 | 5
Not completed — Subject withdrawn due to exclusion criteria (bilateral knee) | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) is a subset of the Safety Population (SAF) that included enrolled participants with data collected for at least one post-operative assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA) | Total
Number analyzed (Participants) | 55 | 71 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (7.3) | 65.0 (9.9) | 64.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 38 | 67
  Male | 26 | 33 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White Caucasian | 51 | 61 | 112
  Race: Black or Arican American | 2 | 4 | 6
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian Indian | 2 | 5 | 7
  Race: Chinese | 0 | 0 | 0
  Race: Japanese | 0 | 0 | 0
  Race: Filipino | 0 | 0 | 0
  Race: Korean | 0 | 0 | 0
  Race: Vietnamese | 0 | 1 | 1
  Race: Other Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 39 | 71
  United Kingdom | 6 | 6 | 12
  Germany | 15 | 21 | 36
  India | 2 | 5 | 7
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 168.6 (11.0) | 170.2 (10.4) | 169.5 (10.6)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 86.4 (16.6) | 87.7 (16.9) | 87.1 (16.7)
Body Mass Index (BMI) [Count of Participants; unit: Participants] — Body Mass Index (BMI) for participants was categorized as one of the following:
  * Underweight (BMI < 18.5)
  * Healthy weight (BMI 18.5 to < 25)
  * Overweight (BMI 25 to < 30)
  * Class 1 obesity (BMI 30 to < 35)
  * Class 2 obesity (BMI 35 to <40)
  * Class 3 obesity (BMI 40 or over)
  Participants
    Underweight (BMI < 18.5) | 0 | 1 | 1
    Healthy weight (BMI 18.5 to < 25) | 7 | 6 | 13
    Overweight (BMI 25 to < 30) | 22 | 29 | 51
    Class 1 obesity (BMI 30 to < 35) | 16 | 22 | 38
    Class 2 obesity (BMI 35 to <40) | 10 | 13 | 23
    Class 3 obesity (BMI 40 or over) | 0 | 0 | 0
Primary Diagnosis [Count of Participants; unit: Participants] — Primary diagnosis for participants was categorized as either osteoarthritis or rheumatoid arthritis
  Participants
    Osteoarthritis | 55 | 69 | 124
    Rheumatoid arthritis | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Leg Alignment
Description: The number of participants with knees achieving post-operative leg alignment was taken by radiographic assessment at 6 weeks. Post-operative leg alignment was achieved when the deviation from the participant specific target did not exceed ±3 degrees. Participants achieving post-operative leg alignment were categorized by the following procedure types: Unicondylar Knee Arthroplasty (UKA), Total Knee Arthroplasty (TKA), and overall (i.e., both procedures).
Time Frame: 6 weeks
Population: Full analysis set included participants with at least one post-operative assessment up to the primary completion date with data collected for the time frame, procedure type, and outcome indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | CORI Robotics
Number analyzed (Participants) | 109
Participants
  Unicondylar Knee Arthroplasty (UKA): number analyzed (Participants) | 47
  Unicondylar Knee Arthroplasty (UKA) | 42
  Total Knee Arthroplasty (TKA): number analyzed (Participants) | 62
  Total Knee Arthroplasty (TKA) | 55
  Overall | 97

2. Primary Outcome: Percentage of Knees Achieving Post-Operative Leg Alignment
Description: The percentage of knees achieving post-operative leg alignment taken by radiographic assessment at 6 weeks. Post-operative leg alignment was achieved when the deviation from the participant specific target did not exceed ±3 degrees. Percentage of knees achieving post-operative leg alignment were categorized by the following procedure types: Unicondylar Knee Arthroplasty (UKA), Total Knee Arthroplasty (TKA), and overall (i.e., both procedures).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of knees
Units Other Than Participants: knees
Arm/Group | CORI Robotics
Number analyzed (Participants) | 109
Number analyzed (knees) | 109
percentage of knees
  Unicondylar Knee Arthroplasty (UKA): number analyzed (Participants) | 47
  Unicondylar Knee Arthroplasty (UKA): number analyzed (knees) | 47
  Unicondylar Knee Arthroplasty (UKA) | 89.36 [76.9 to 96.45]
  Total Knee Arthroplasty (TKA): number analyzed (Participants) | 62
  Total Knee Arthroplasty (TKA): number analyzed (knees) | 62
  Total Knee Arthroplasty (TKA) | 88.71 [78.11 to 95.34]
  Overall | 88.99 [81.56 to 94.18]

3. Secondary Outcome: Component Alignment: Femoral Antero-Posterior (A/P) Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. From the A/P radiograph, the femoral flexion angle is to be obtained using standard radiographic tools. Femoral flexion angle is defined as the angle formed between a line across the base of the femoral condyles and a line that is centered along the femoral canal.
Time Frame: 6 weeks
Population: Full analysis set (FAS) included enrolled participants that had at least one post-operative assessment with data collected for the time frame specified.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 47 | 64
degrees | 94.0 (4.5) | 92.4 (4.3)

4. Secondary Outcome: Component Alignment: Tibial Antero-Posterior (A/P) Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. From the A/P radiograph, the tibial angle denotes the angle formed on the medial side of the knee from intersecting lines parallel to the tibial base plate and a line drawn parallel to the tibial canal.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 47 | 64
degrees | 88.6 (2.9) | 89.5 (1.9)

5. Secondary Outcome: Component Alignment: Total Valgus Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. The total valgus angle is the sum of the femoral flexion angle and the tibial angle.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 47 | 64
degrees | 182.6 (6.0) | 181.9 (5.1)

6. Secondary Outcome: Component Alignment: Femoral Flexion Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. The lateral view femoral flexion angle is obtained from the intersection of a line from the center of the femoral implant to the top of the femur with a line through the femoral canal. The angle is measured on the proximal side of the intersection.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 45 | 63
degrees | 3.4 (4.1) | 3.3 (1.8)

7. Secondary Outcome: Component Alignment: Tibial Lateral Angle
Description: Component alignment assessed on long leg standing antero-posterior (A/P) X-rays and standard non weight bearing lateral X-rays taken 6 weeks after surgery. The lateral view tibial angle is the angle obtained from the intersection of a line drawn parallel to the bottom of the tibial base insert and a line through the center of the tibial base and the tibial canal.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 45 | 63
degrees | 84.6 (12.9) | 83.8 (18.0)

8. Secondary Outcome: Radiographic Assessment: Radiographic Findings
Description: Radiographic assessment on antero-posterior (A/P) and lateral (L) views were performed to identify radiographic findings for the presence of radiolucent lines, osteolysis and implant migration. The number of participants with radiographic findings were categorized as one of the following:
  * Yes
  * No
  * Missing
Time Frame: 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 45 | 61
Participants
  Yes | 0 | 0
  Missing | 3 | 5
  No | 42 | 56

9. Secondary Outcome: 2011 Knee Society Score (KSS): Objective Score
Description: The 2011 Knee Society Score Objective score is completed by the surgeon and assesses the condition of the knee based on factors like pain, alignment, ligament stability, and range of motion. The Objective score ranges from 0 to 100, with a higher score indicating better knee function (i.e., a better outcome).
Time Frame: Pre-op, 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 54 | 61
score on a scale
  Pre-Op | 20.9 (15.8) | 19.3 (15.7)
  6 weeks: number analyzed (Participants) | 49 | 61
  6 weeks | 44.7 (18.9) | 44.1 (18.2)
  6 months: number analyzed (Participants) | 34 | 30
  6 months | 51.9 (18.8) | 46.5 (16.4)
  12 months: number analyzed (Participants) | 41 | 53
  12 months | 51.9 (18.9) | 46.5 (17.0)

10. Secondary Outcome: 2011 Knee Society Score (KSS): Function Score
Description: The 2011 Knee Society Score Function assesses the participant's ability to perform daily activities and is a component of the overall KSS evaluation. The Function score ranges from 0 to 100, with a higher score indicating better function (i.e., a better outcome).
Time Frame: Pre-op, 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 32 | 37
score on a scale
  Pre-Op | 43.6 (10.9) | 45.0 (11.3)
  6 weeks: number analyzed (Participants) | 18 | 25
  6 weeks | 59.0 (13.5) | 54.1 (15.7)
  6 months: number analyzed (Participants) | 27 | 29
  6 months | 66.5 (13.9) | 65.9 (12.8)
  12 months: number analyzed (Participants) | 24 | 29
  12 months | 73.7 (9.0) | 69.2 (13.8)

11. Secondary Outcome: 2011 Knee Society Score (KSS): Satisfaction Score
Description: The 2011 Knee Society Score Satisfaction score is a five question 40-point scale completed by the participant. The Satisfaction score ranges from 0 to 40, with a higher score indicating greater satisfaction (i.e., a better outcome).
Time Frame: Pre-op, 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 55 | 71
score on a scale
  Pre-Op | 13.8 (6.9) | 12.8 (7.1)
  6 weeks: number analyzed (Participants) | 51 | 65
  6 weeks | 25.6 (8.0) | 23.7 (7.7)
  6 months: number analyzed (Participants) | 48 | 61
  6 months | 31.0 (9.5) | 29.5 (9.2)
  12 months: number analyzed (Participants) | 44 | 61
  12 months | 33.9 (7.7) | 30.5 (9.3)

12. Secondary Outcome: Oxford Knee Score (OKS)
Description: The Oxford Knee Score (OKS) specifically assesses the patient's perspective following knee arthroplasty surgery to indicate knee function. Total overall scores range from 0 to 48. A score of 0 is the worst possible outcome while a score of 48 indicates the best possible outcome.
Time Frame: Pre-op, 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 55 | 71
score on a scale
  Pre-op | 23.2 (7.5) | 21.8 (7.8)
  6 weeks: number analyzed (Participants) | 49 | 65
  6 weeks | 30.6 (7.9) | 27.0 (7.2)
  6 months: number analyzed (Participants) | 48 | 61
  6 months | 39.3 (8.5) | 37.0 (8.4)
  12 months: number analyzed (Participants) | 42 | 61
  12 months | 41.8 (7.5) | 38.4 (8.0)

13. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The forgotten Joint Score (FJS) consisted of 12 questions with responses recorded using a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores were summed and linearly transformed to a 0 to 100 scale and then reversed with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living. A score of 100 is the best possible outcome (i.e., a high score indicated a better outcome).
Time Frame: 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 47 | 62
score on a scale
  6 weeks | 35.0 (26.6) | 27.5 (24.4)
  6 months: number analyzed (Participants) | 45 | 60
  6 months | 57.7 (32.4) | 46.0 (31.8)
  12 months: number analyzed (Participants) | 43 | 60
  12 months | 68.0 (27.9) | 51.2 (36.0)

14. Secondary Outcome: Five-level EuroQol Five-dimensional (EQ-5D-5L) Visual Analogue Scale (VAS) Score
Description: The EQ-5D-5L is composed of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The EQ VAS score uses a scale from 0 to 100, with 0 indicating 'the worst health you can imagine' (i.e., a worse outcome) and 100 indicating 'the best health you can imagine' (i.e., a better outcome).
Time Frame: Pre-op, 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 55 | 67
score on a scale
  Pre-op | 69.2 (18.27) | 66.27 (19.48)
  6 weeks: number analyzed (Participants) | 53 | 63
  6 weeks | 77.04 (18.37) | 76.13 (18.24)
  6 months: number analyzed (Participants) | 48 | 60
  6 months | 79.08 (16.81) | 78.75 (16.94)
  12 months: number analyzed (Participants) | 45 | 61
  12 months | 84.27 (13.76) | 81.0 (15.25)

15. Secondary Outcome: Five-level EuroQol Five-dimensional (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is composed of the EQ-5D-5L descriptive system (i.e., index score) and the EQ Visual Analogue scale (EQ VAS). The descriptive system is a health-related quality of life score that comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. A score of 1 indicates perfect health-related quality of life and 0 indicates no health-related quality of life (i.e., a higher score is a better outcome). Index scores cannot be greater than 1 but could be less than 0.
Time Frame: Pre-op, 6 weeks, 6 months and 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
Number analyzed (Participants) | 55 | 67
score on a scale
  Pre-op | 0.63 (0.19) | 0.58 (0.21)
  6 weeks: number analyzed (Participants) | 53 | 63
  6 weeks | 0.79 (0.13) | 0.75 (0.14)
  6 months: number analyzed (Participants) | 48 | 59
  6 months | 0.84 (0.14) | 0.82 (0.12)
  12 months: number analyzed (Participants) | 45 | 61
  12 months | 0.88 (0.12) | 0.85 (0.12)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of enrollment to study completion, approximately 12 months.
Description: The Safety Population (SAF) included enrolled participants that were treated for UKA or TKA using CORI™ Robotics with data collected.
Arm/Group | CORI™ in Unicondylar Knee Arthroplasty (UKA) | CORI™ in Total Knee Arthroplasty (TKA)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/71
Serious Adverse Events (participants affected / at risk) | 2/55 | 10/71
Other Adverse Events (participants affected / at risk) | 17/55 | 26/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CORI™ in Unicondylar Knee Arthroplasty (UKA) (N=55) | CORI™ in Total Knee Arthroplasty (TKA) (N=71)
UNSPECIFIED GASTROINTESTINAL PROBLEM (Gastrointestinal disorders) | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
INTERVERTEBRAL DISC COMPRESSION OR PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
LOSS OF RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 1 | 3
JOINT CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
FIBROSIS (General disorders) | 0 | 2
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CORI™ in Unicondylar Knee Arthroplasty (UKA) (N=55) | CORI™ in Total Knee Arthroplasty (TKA) (N=71)
NERVOUS SYSTEM INJURY (Nervous system disorders) | 1 | 0
NUMBNESS (Nervous system disorders) | 0 | 1
PERIPHERAL NERVOUS INJURY (Nervous system disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1
UNSPECIFIED GASTROINTESTINAL PROBLEM (Gastrointestinal disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 3
JOINT LAXITY (Musculoskeletal and connective tissue disorders) | 1 | 0
LOSS OF RANGE OF MOTION (Musculoskeletal and connective tissue disorders) | 0 | 1
UNSPECIFIED MUSCULOSKELETAL PROBLEM (Musculoskeletal and connective tissue disorders) | 0 | 1
NODULE (Musculoskeletal and connective tissue disorders) | 0 | 1
BACTERIAL INFECTION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UNSPECIFIED INFECTION (Infections and infestations) | 1 | 0
FALL (Infections and infestations) | 3 | 2
AMBULATION DIFFICULTIES (Injury, poisoning and procedural complications) | 0 | 1
INFLAMMATION (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN (General disorders) | 7 | 7
SWELLING/ EDEMA (General disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT04786119/Prot_SAP_000.pdf